CLINICAL TRIAL: NCT01362712
Title: An Exploratory, Phase I, Open Label, Multi-Center, Non-randomized Study of [F18]CP-18 PET in Normal and Breast Cancer Subjects
Brief Title: Exploratory, Phase I,Open Label,Non-randomized Study of [F18]CP-18 PET in Normal and Breast Cancer Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to enroll breast cancer patients with current I/E criteria.
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP-18 100
Record Dates: First submitted 2011-05-13; First posted 2011-05-30 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; radiotherapy; chemoradiotherapy; radiation; chemoradiation; [F-18]
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: [F18]CP-18 Injection — Normal volunteers dose will not exceed 20 mCi. For cancer subjects, the dose will be closer to 10 mCi.
  Other Names: [F18]CP-18

SUMMARY:
This trial will be the first trial for the IP, [F-18]CP-18, and will be conducted as an exploratory Phase I trial designed to collect information as this IP is administered and evaluated for the first time in humans. The trial will evaluate safety, biodistribution and dosimetry data in normal subjects and the trial will evaluate safety, biodistribution and tumor to background imaging data, and correlate image data with caspase 3 activity level on a surgical specimen analyzed by immunohistochemistry in the cancer subjects. All study results will be evaluated and analyzed in order to consider the design for future clinical trials. The information collected under this exploratory, Phase I study will not be used for diagnostic purposes, to assess the subject's response to therapy, or for clinical management of the subject.

DETAILED DESCRIPTION:
The Sponsor intends to conduct this exploratory investigation of [F-18]CP-18 in human subjects. In this study of [F-18]CP-18, it is intended to assess its biodistribution, PET scan resolution, signal to background ratio in tumor, and any adverse events. This exploratory Phase I study will be used to obtain the necessary safety and dosimetry data in normal subjects and to collect drug biodistribution data, and tumor to background imaging data in breast cancer subjects. The information collected from this study will not be used for diagnostic purposes, to assess the subject's response to therapy, or for clinical management of the subject.

ELIGIBILITY:
Inclusion Criteria:

For Normal Volunteers

* Subject is a female or male of any race / ethnicity between 21 to 75 years old at the time of the investigational product administration
* Subject or subject's legally acceptable representative provides written informed consent
* Subject is capable of complying with study procedures
* Subject must have renal functions values as defined by laboratory results within the following ranges:
* Serum creatinine ≤ 2x institutional upper limits of normal

For Cancer Patients

* Patient is a female or male of any race / ethnicity between 21 to 75 years old at the time of the investigational product administration
* Patients or subject's legally acceptable representative provides written informed consent
* Patient is capable of complying with study procedures
* Patient must have renal functions values as defined by laboratory results within the following ranges:
* Serum creatinine ≤ 2x institutional upper limits of normal
* BUN < 2X institutional upper limits of normal
* Patient must have a confirmed diagnosis of stage IIB/IIIA/IIIB, locally advanced breast cancer
* Patient has been or will be scheduled for the surgical resection of tumor(s) after undergoing neoadjuvant treatment and within approximately 7 days following the [F-18]CP-18 PET/CT scan
* Patient has an adequate size breast tumor (≥1.0 cm) that should be amenable to imaging
* Patient's tumor tissue is obtainable following surgery in order to perform immunohistochemistry staining using caspase 3 and/or other apoptosis biomarkers
* Patient must have a previous baseline (pre-neoadjuvant treatment) diagnostic imaging exam including but not limited to MRI, CT, mammography, or [F-18] FDG PET/CT scan that identifies breast tumor location

Exclusion Criteria:

For Normal Volunteers

* Subject is nursing
* Subject is pregnant
* Subject has been involved in an investigative, radioactive research procedure within the past 14 days
* Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete data or data quality

For Cancer Patients

* Subject is nursing
* Subject is pregnant
* Subject has been involved in an investigative, radioactive research procedure within the past 14 days
* Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete data or data quality
* Patient tumor tissue(s) is not obtainable after tumor resection for caspase 3 and/or other biomarker immunohistochemistry assays
* Patient has had or will have treatment intervention(s) between the [F-18]CP-18 PET/CT scan and tumor resection
* Patient has a history or current evidence of any condition, therapy, lab abnormality that, in the opinion of the study investigator or treating physicians might confound the results of the study or poses an additional risk to the patients by their participation in the study

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To collect biodistribution, dosimetry and metabolite profile of [F-18]CP-18 from normal subjects | Visit 2 and Visit 3

SECONDARY OUTCOMES:
To collect pre-dose and post-dose parameters of vital signs, ECG and CBC and clinical chemistry data along with monitoring any adverse events of the IP from normal and cancer subjects. | Visit 2 and Visit 3

CONTACTS AND LOCATIONS:
Overall Officials: Edward Aten, MD, Study Director — President, Certus International Inc. Medical Monitor; Michael Yu, MD, Principal Investigator — FCCC
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Doss M, Kolb HC, Walsh JC, Mocharla V, Fan H, Chaudhary A, Zhu Z, Alpaugh RK, Lango MN, Yu JQ. Biodistribution and radiation dosimetry of 18F-CP-18, a potential apoptosis imaging agent, as determined from PET/CT scans in healthy volunteers. J Nucl Med. 2013 Dec;54(12):2087-92. doi: 10.2967/jnumed.113.119800. Epub 2013 Oct 17. PMID 24136934